CLINICAL TRIAL: NCT03578146
Title: A Randomized, Double-Blind, Vehicle-Controlled Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously Administered PRT064445 After Dosing to Steady State With One of Four Direct/Indirect fXa Inhibitors in Healthy Volunteers
Brief Title: Phase 2 Healthy Volunteer Study to Evaluate the Ability of PRT064445 to Reverse the Effects of Several Blood Thinner Drugs on Laboratory Tests (Module 2 of 4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-502 Module 2
Record Dates: First submitted 2018-05-15; First posted 2018-07-06 (Actual); Results first posted 2018-09-05 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PRT064445; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: This study has four modules with a total of 21 cohorts, each module was reported and submitted separately.
  Module 1, NCT01758432 (54 subjects with 7 cohorts including placebo); Module 2, NCT03578146 (48 subjects with 6 cohorts including placebo); Module 3, NCT03551730 (27 subjects with 4 cohorts including placebo); Module 4, NCT03551743 (28 subjects with 4 cohorts including placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Module 2 (210 mg) (Experimental): 210 mg andexanet IV bolus administered over 7 minutes (~30 mg/min)
  Interventions: Combination Product: PRT064445/Rivaroxaban; Combination Product: Placebo/Rivaroxaban
- Module 2 (420 mg) (Experimental): 420 mg andexanet IV bolus administered over 14 minutes (~30 mg/min)
  Interventions: Combination Product: PRT064445/Rivaroxaban; Combination Product: Placebo/Rivaroxaban
- Module 2 (600 mg) (Experimental): 600 mg andexanet IV bolus administered over 20 minutes (~30 mg/min)
  Interventions: Combination Product: PRT064445/Rivaroxaban; Combination Product: Placebo/Rivaroxaban
- Module 2 (720 mg bolus + 240 mg infusion) (Experimental): 720 mg IV bolus administered over 24 minutes [~30 mg/min] followed by 240 mg continuous IV infusion [4 mg/min over 60 min)
  Interventions: Combination Product: PRT064445/Rivaroxaban; Combination Product: Placebo/Rivaroxaban
- Module 2 (800 mg bolus + 960 mg infusion) (Experimental): 800 mg IV bolus administered over 26.7 minutes [~30 mg/min] followed by 960 mg continuous IV infusion [8 mg/min over 120 min]
  Interventions: Combination Product: PRT064445/Rivaroxaban; Combination Product: Placebo/Rivaroxaban
- Module 2 Placebo (Experimental): Placebo administered intravenously (IV) as a bolus or a bolus followed by continuous fusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: PRT064445/Rivaroxaban
  Other Names: Andexanet
  Arms: Module 2 (210 mg); Module 2 (420 mg); Module 2 (600 mg); Module 2 (720 mg bolus + 240 mg infusion); Module 2 (800 mg bolus + 960 mg infusion)
Combination Product: Placebo/Rivaroxaban
  Arms: Module 2 (210 mg); Module 2 (420 mg); Module 2 (600 mg); Module 2 (720 mg bolus + 240 mg infusion); Module 2 (800 mg bolus + 960 mg infusion)
Drug: Placebo
  Arms: Module 2 Placebo

SUMMARY:
The purpose of this study is to evaluate the ability of PRT064445 to reverse the effects of several blood thinner drugs on laboratory tests. The study also is evaluating the blood levels of PRT064445 given at different doses.

DETAILED DESCRIPTION:
A randomized, double-blind, vehicle-controlled study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of intravenously administered PRT064445 after dosing to steady state with one of four direct/indirect factor Xa (fXa) inhibitors in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between the ages of 18 and 45 years old

Exclusion Criteria:

* History (including family history) or symptoms of, or risk factors for bleeding
* History (including family history) of or risk factors for a hypercoagulable or thrombotic condition
* Absolute/relative contraindication to anticoagulation or treatment with specific anticoagulants
* History of major surgery, severe trauma or bone fracture within 3 months prior to dosing; or planned surgery within 1 month after dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

REFERENCES:
- [Derived] Lu G, Conley PB, Leeds JM, Karbarz MJ, Levy GG, Mathur VS, Castillo J, Crowther M, Curnutte JT. A phase 2 PK/PD study of andexanet alfa for reversal of rivaroxaban and edoxaban anticoagulation in healthy volunteers. Blood Adv. 2020 Feb 25;4(4):728-739. doi: 10.1182/bloodadvances.2019000885. PMID 32092140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative site in the US between March 2013 through April 2014
Pre-assignment Details: Rivaroxaban was administered orally at 20 mg once daily for 6 days to steady-state in an open label fashion. Subjects were then randomized to receive study treatment (andexanet or placebo) intravenously at different doses/dose regimens on Day 6, all bolus doses administered such that they ended at 3 hours after the last dose of rivaroxaban.
Groups:
- Module 2 Placebo: Placebo administered intravenously (IV) as a bolus or a bolus followed by continuous infusion
Period: Overall Study
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Started | 16 | 6 | 6 | 6 | 6 | 8
Completed | 15 | 5 | 5 | 6 | 6 | 5
Not Completed | 1 | 1 | 1 | 0 | 0 | 3
Not completed — Did Not Receive Treatment | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 48 subjects were enrolled in this study. Three subjects received rivaroxaban but were discontinued prior to receiving andexanet/placebo due to problems with the infusion pumps observed in prior subjects in the cohort and these subjects were replaced.
Groups:
- Total: Total of all reporting groups
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion) | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (6.69) | 35.7 (3.33) | 35.7 (9.07) | 34.2 (7.25) | 35.2 (5.04) | 32.9 (8.10) | 35.8 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 4 | 0 | 1 | 9
  Male | 13 | 6 | 5 | 2 | 6 | 7 | 39

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percent Change From Baseline in Anti-fXa Activity at 2 Mins Following Andexanet/Placebo Administration
Description: Anti-fXa activity was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Anti-fXa activity was measured using a commercial kit (Coamatic Heparin-82 33 9363, DiaPharma)
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 45 subjects who received andexanet or placebo were included in the pharmacodynamics (PD) analysis
Measure: Mean (Standard Deviation); unit: Percent change in anti-fXa activity
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
Percent change in anti-fXa activity | 22.37 (42.247) | -18.09 (23.922) | -50.59 (22.056) | -75.26 (19.072) | -88.91 (6.098) | -92.72 (3.084)
Statistical Analysis 1: Comparison: Module 2 Placebo vs Module 2 (210 mg); Test type: Superiority; p = 0.0121, ANCOVA; Least Squares Means (Difference) = -73.14
Statistical Analysis 2: Comparison: Module 2 Placebo vs Module 2 (420 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -153.99
Statistical Analysis 3: Comparison: Module 2 Placebo vs Module 2 (600 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -189.57
Statistical Analysis 4: Comparison: Module 2 Placebo vs Module 2 (720 mg Bolus + 240 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -239.3
Statistical Analysis 5: Comparison: Module 2 Placebo vs Module 2 (800 mg Bolus + 960 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -231.12

2. Secondary Outcome: Efficacy: Percent Change From Baseline in Thrombin Generation at 2 Mins Following Andexanet/Placebo Administration
Description: Thrombin generation was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Thrombin generation was measured using a TF-initiated thrombin generation assay.
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 45 subjects who received andexanet or placebo were included in the PD analysis
Measure: Mean (Standard Deviation); unit: Percent change in thrombin generation
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
Percent change in thrombin generation | 14.00 (29.267) | 107.47 (48.977) | 167.67 (36.568) | 246.02 (135.387) | 513.85 (285.992) | 559.14 (288.258)
Statistical Analysis 1: Comparison: Module 2 Placebo vs Module 2 (210 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 52837.94
Statistical Analysis 2: Comparison: Module 2 Placebo vs Module 2 (420 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 110388.3
Statistical Analysis 3: Comparison: Module 2 Placebo vs Module 2 (600 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 163880.7
Statistical Analysis 4: Comparison: Module 2 Placebo vs Module 2 (720 mg Bolus + 240 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 263236.5
Statistical Analysis 5: Comparison: Module 2 Placebo vs Module 2 (800 mg Bolus + 960 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 270297.2

3. Secondary Outcome: Efficacy: Percent Change From Baseline in Unbound Rivaroaxaban Plasma Concentration at 2 Mins Following Andexanet/Placebo Administration
Description: Unbound rivaroxaban concentrations was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Unbound plasma concentrations for rivaroxaban were determined by a rapid equilibrium dialysis method followed by Liquid Chromatography-Mass Spectometry assay.
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 45 subjects who received rivaroxaban were included in the rivaroxaban pharmacokinetics (PK) analysis
Measure: Mean (Standard Deviation); unit: Percent change in unbound apixaban conc.
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
Percent change in unbound apixaban conc. | -11 (11) | 34 (22) | 52 (18) | 75 (16) | 67 (24) | 80 (12)
Statistical Analysis 1: Comparison: Module 2 Placebo vs Module 2 (210 mg); Test type: Superiority; p = 0.002, ANCOVA; Least Squares Means (Difference) = -9.91
Statistical Analysis 2: Comparison: Module 2 Placebo vs Module 2 (420 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -15.06
Statistical Analysis 3: Comparison: Module 2 Placebo vs Module 2 (600 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -17.53
Statistical Analysis 4: Comparison: Module 2 Placebo vs Module 2 (720 mg Bolus + 240 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -17.05
Statistical Analysis 5: Comparison: Module 2 Placebo vs Module 2 (800 mg Bolus + 960 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -19.33

4. Secondary Outcome: Andexanet Maximum Observed Plasma Concentration (Cmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay.
Time Frame: Blood was collected at predose, 0.033, 0.2, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5.5, 6.5, 7.5, 8.5 and 14.5 hours postdose.
Population: 30 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
ng/mL | NA (NA) — Andexanet was not administered (placebo group) | 50400 (12100) | 105000 (28500) | 110000 (7070) | 123000 (28900) | 161000 (40400)

5. Secondary Outcome: Andexanet Area Under the Drug Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf )
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. AUC0-inf was calculated using a non-compartmental approach
Time Frame: as for outcome 4
Population: 30 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | NA (NA) — Andexanet was not administered (placebo group) | 51400 (7520) | 111000 (35900) | 133000 (11500) | 216000 (41300) | 429000 (85300)

6. Secondary Outcome: Andexanet Time of Maximum Observed Plasma Concentration (Tmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Tmax was taken directly from the raw data.
Time Frame: as for outcome 4
Population: 30 subjects who received andexanet were included in the andexanet PK analysis
Measure: Median (Full Range); unit: hr
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
hr | NA [NA to NA] — Andexanet was not administered (placebo group) | 0.17 [0.16 to 0.41] | 0.36 [0.29 to 0.52] | 0.51 [0.39 to 0.83] | 0.56 [0.44 to 0.70] | 0.52 [0.49 to 0.73]

7. Secondary Outcome: Andexanet Apparent Terminal Elimination Half-life (t1/2)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. t1/2 was determined by linear regression of the log concentration on the terminal portion of the plasma concentration-time curve.
Time Frame: as for outcome 4
Population: 30 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
hr | NA (NA) — Andexanet was not administered (placebo group) | 4.97 (0.74) | 3.91 (0.43) | 4.54 (1.65) | 6.47 (3.59) | 4.45 (0.58)

8. Secondary Outcome: Andexanet Total Systemic Clearance (CL)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. CL was calculated using a non-compartmental approach, calculated as Dose/AUC0-inf
Time Frame: as for outcome 4
Population: 30 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
L/hr | NA (NA) — Andexanet was not administered (placebo group) | 4.15 (0.556) | 4.18 (1.51) | 4.53 (0.399) | 4.58 (0.837) | 4.23 (0.808)

9. Secondary Outcome: Andexanet Total Volume of Distribution (Vss)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Vss was calculated using a non-compartmental approach.
Time Frame: as for outcome 4
Population: 30 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6
L | NA (NA) — Andexanet was not administered (placebo group) | 5.23 (1.09) | 4.65 (1.69) | 5.39 (0.546) | 4.17 (0.797) | 3.34 (1.20)

ADVERSE EVENTS:
Time Frame: ~7 weeks
Description: Only subjects who received at least one dose of study drug were included in the safety analysis.
Arm/Group | Module 2 Placebo | Module 2 (210 mg) | Module 2 (420 mg) | Module 2 (600 mg) | Module 2 (720 mg Bolus + 240 mg Infusion) | Module 2 (800 mg Bolus + 960 mg Infusion)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 12/15 | 4/6 | 3/6 | 5/6 | 5/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Module 2 Placebo (N=15) | Module 2 (210 mg) (N=6) | Module 2 (420 mg) (N=6) | Module 2 (600 mg) (N=6) | Module 2 (720 mg Bolus + 240 mg Infusion) (N=6) | Module 2 (800 mg Bolus + 960 mg Infusion) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site reaction (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Vessel puncture site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2 | 3 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0 | 2 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 2 | 0 | 1 | 2 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 1 | 2 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tunnel vision (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Conducted in healthy volunteers at Clinical Research Organization.